## The GlaxoSmithKline group of companies

| Division | · | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan (RAP) for 201023: A Phase II, global, randomized study to evaluate the efficacy and safety of Danirixin (GSK1325756) co-administered with a standard-of-care antiviral (oseltamivir), in the treatment of adults hospitalized with influenza |
|---|---|---|
| <b>Compound Number</b> | : | GSK1325756 |
| <b>Effective Date</b> | : | 05-SEP-2017 |

## **Description:**

- 1. The purpose of this RAP is to describe the planned analyses and output to be included in the Synoptic Report for study 201023. This document contains the RAP Amendment 01.
- 2. This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

### **Author's Name and Functional Area:**

| PPD | |
|-------------------------------------|-------------------|
| Director (Sta | tistics, PAREXEL) |
| PPD | |
| Director (Clinical Statistics, GSK) | |

## **Electronically Approved by:**

| PPD | | |
|------------------------|-------------|--------|
| Director (Clinical Sta | 05-SEP-2017 | |
| Manager (Programmi | ng, GSK) | 32 231 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | ORTING & ANALYSIS PLAN SYNOPSIS | 5 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses. | |
| | ۷.٦. | Oldifoliodi Frypotriosos | |
| 3. | PLAN | INED ANALYSES | 9 |
| | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | |
| | | , | |
| 4. | ANAL' | YSIS POPULATIONS | 10 |
| | 4.1. | Protocol Deviations | 10 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | VENTIONS | 11 |
| 6. | | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | 12 |
| _ | DD114 | ADV OTATIOTICAL ANALYOFO | 4.4 |
| 7. | | ARY STATISTICAL ANALYSES | |
| | 7.1. | ,, | |
| | | 7.1.1. Overview of Planned Efficacy Analyses | |
| | | 7.1.2. Planned Efficacy Statistical Analyses | 14 |
| 8. | SECO | ONDARY STATISTICAL ANALYSES | 16 |
| Ο. | 8.1. | Efficacy Analyses | |
| | 0.1. | 8.1.1. Overview of Planned Efficacy Analyses | |
| | 8.2. | Safety Analyses | |
| | 0.2. | 8.2.1. Overview of Planned Adverse Events Analyses | |
| | | 8.2.2. Overview of Planned Clinical Laboratory Analyses | |
| | | 8.2.3. Overview of Planned Other Safety Analyses | |
| | 8.3. | Pharmacokinetic Analyses | 20 |
| | 0.0. | Pharmacokinetic Analyses | 20 |
| | | 8.3.2. Drug Concentration Measures | |
| | | 8.3.3. Pharmacokinetic Parameters | |
| | | 8.3.3.1. Deriving Pharmacokinetic Parameters | |
| | | 8.3.3.2. Statistical Analysis of Pharmacokinetic | |
| | | Parameters | 21 |
| | | 8.3.4. Population Pharmacokinetic (PopPK) Analyses | |
| | 8.4. | Biomarker Analyses | |
| | | 8.4.1. Overview of Planned Biomarker Analyses | |
| | 8.5. | Pharmacodynamic / Biomarker Statistical Analyses | |
| | | 8.5.1. Overview of Planned Pharmacodynamic / Biomarker | |
| | | Analyses | <mark>22</mark> |
| | 8.6. | Pharmacokinetic / Pharmacodynamic Analyses | |
| | 8.7. | Health Outcome Analyses | 23 |
| | | 8.7.1. Overview of Planned Health Outcome Analyses | |


| 201023 |
|--------|
| 201023 |

| 9. | <b>VIROL</b> | OGY ANA | LYSES | | 23 |
|---|---|---|---|---|---|
| | 9.1. | Overview | of Planned | l Virology Analyses | 23 |
| | 9.2. | Planned \ | /irology Sta | atistical Analyses | 24 |
| | | | | • | |
| 10. | REFE | RENCES | | | 26 |
| 11. | | | | | 27 |
| | 11.1. | Protocol F | Population | I Deviation Management and Definitions for Per | 28 |
| | 11.2. | <b>Appendix</b> | 2: Time & | Events | 28 |
| | | | | efined Time & Events | |
| | 11.3. | | | ment Windows | |
| | 11.4. | | | ent States and Phases | |
| | | | | Phases | |
| | | | | States | 32 |
| | | | | Treatment States for Concomitant Medications | |
| | | | | Data | |
| | 44.5 | | | Treatment States for AE Data | |
| | 11.5. | | | splay Standards & Handling Conventions | |
| | | 11.5.1. | Study Trea | Itment & Sub-group Display Descriptors | 33 |
| | | | | efinition & Derivations | |
| | | | | Baseline Definitions | 34 |
| | | | 11.3.2.2. | Derivations and Handling of Missing Baseline Data | 3/1 |
| | | 11.5.3. | | Process & Standards | |
| | 11.6. | | | and Transformed Data | |
| | 11.0. | | | and Transformed Data | |
| | | | | ulation | |
| | | | 11.6.5.1. | Biomarkers and Source | 39 |
| | | 11.6.6. | Health Out | comes | 40 |
| | 11.7. | <b>Appendix</b> | 7: Prematu | ure Withdrawals & Handling of Missing Data | 42 |
| | | 11.7.1. | Premature | Withdrawals | 42 |
| | | | | f Missing Data | |
| | | | | Handling of Missing Dates | |
| | | | | Handling of Partial Dates | 43 |
| | | | | Handling of Missing Data for Statistical | |
| | | | | Analysis | 43 |
| | 11.8. | Appendix | 8: Values | of Potential Clinical Importance | 43 |
| | | | | Values | |
| | 44.0 | | | | |
| | 11.9. | | | ation of Covariates, Subgroups & Other Strata | |
| | 11 10 | | | on of Covariates, Subgroups & Other Strata | |
| | 11.10. | | | e Comparisons & Multiplicity | |
| | 11 11 | | | f Multiple Comparisons & Multiplicity Checking and Diagnostics for Statistical | 44 |
| | 11.11. | | | Statistical | 41 |
| | | 11 11 1 | Statistical A | Analysis Assumptions | <u>++</u> |
| | 11 12 | | | eviations & Trade Marks | |
| | | | , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | |


201023

| | 11.12.1. | Abbreviations | .44 |
|--------|----------|--------------------------------------------|-----|
| | 11.12.2. | Trademarks | .44 |
| 11.13. | Appendix | c 13: List of Data Displays | .45 |
| | 11.13.1. | Data Display Numbering | .45 |
| | 11.13.2. | Mock Example Shell Referencing | .45 |
| | 11.13.3. | Deliverable [Priority] | .46 |
| | 11.13.4. | Study Population Tables | .47 |
| | | Efficacy Tables | |
| | 11.13.6. | Efficacy Figures | .49 |
| | 11.13.7. | Safety Tables | .51 |
| | 11.13.8. | Safety Figures | .53 |
| | 11.13.9. | Pharmacokinetic Tables | .54 |
| | 11.13.10 | .Pharmacokinetic Figures | .55 |
| | 11.13.11 | .Biomarker Figures | .55 |
| | 11.13.12 | .Pharmacodynamic / Biomarker Figures | .57 |
| | 11.13.13 | .Pharmacokinetic / Pharmacodynamic Tables | .59 |
| | 11.13.14 | .Pharmacokinetic / Pharmacodynamic Figures | .59 |
| | 11.13.15 | .Health Outcome Tables | .59 |
| | 11.13.16 | .Virology Tables | .60 |
| | 11.13.17 | .Virology Figures | .60 |
| | | .ICH Listings | |
| | | .Non-ICH Listings | |
| 11.14. | Appendix | 14: Example Mock Shells for Data Displays | .67 |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP describes all the planned analyses and outputs required for the end of study Synoptic Report for study 201023. |
| Protocol | This RAP is based on the original protocol [(Dated: 12/Jul/2016) of study 201023(GSK Document No: 2016N281688_00] and eCRF Version 1 |
| Primary<br>Objective | To assess the efficacy of treatment with IV DNX twice daily given with oral oseltamivir compared to oral oseltamivir twice daily on time to clinical response (TTCR) |
| Primary<br>Endpoint | Time to Clinical Response (composite) • Hospital discharge OR • Normalization of: - Temperature; and - Oxygen status; and - Respiratory status/Heart Rate/SBP(normalization of 2 out of these 3 parameters) |
| Study<br>Design | Phase 2, randomized, double-blind (for IV DNX), placebo-controlled (for IV DNX) 3-arm study in adults to determine the efficacy and safety of IV DNX when coadministered (in all groups) with standard of care antiviral treatment (openlabel oral 75 mg OSV) for patients hospitalized with influenza. |
| | <ul> <li>Enrolled Subjects will be randomized 2:2:1 to 15 mg FBE IV DNX, 50 mg FBE IV DNX, or matching placebo. All subjects will also receive open-label oral OSV, twice daily (given as standard of care).</li> </ul> |
| | Study treatment duration will be for up to 5 days. The investigator may elect to continue treatment with standard of care (OSV) after 5 days of study treatment. |
| | The sample size of 300 was selected based on simulations to achieve at least 80% overall power under assumption of HR =1.5 for 50 mg of DNX FBE and HR =1.2 for 15 mg of DNX FBE and keep type I error less than 10% under no-effect assumption. The study was terminated early after 10 subjects were enrolled. |
| | An Independent Data Monitoring Committee (IDMC) will perform monitoring and reviews of available safety and efficacy data. |
| | All decisions regarding final analysis, as defined in this RAP document, will be made prior to unblinding of the study data. |
| Planned<br>Analyses | The final analysis will occur when both accrual and follow-up are complete for all subjects. |
| Primary<br>Analysis<br>Populations | • 'Influenza Positive Population' (IPP) comprises of all subjects in the ITT-E population with influenza infection (positive influenza PCR or culture at any timepoint) confirmed by central lab testing. |

| Overview | Key Elements of the RAP |
|---|---|
| Hypothesis | No formal hypotheses will be tested and only descriptive summaries will be created for the final analysis. |
| Primary<br>Analyses<br>Secondary<br>Analyses | <ul> <li>Kaplan-Meier estimates for the median of TTCR for each treatment group and 95% confidence interval (CI) will be provided.</li> <li>Median, and 95% CI for time to respiratory response will be provided.</li> <li>Proportion of subjects with clinical response, and improved respiratory status will be summarized.</li> <li>Frequency of antibiotic use</li> <li>Frequency of adverse events (AEs) and serious adverse events (SAEs)</li> <li>Frequency of adverse events of special interest (AESIs)</li> <li>Change from baseline in clinical laboratory evaluations</li> <li>Summarize standard pharmacokinetic parameters for IV DNX (i.e. AUC, Cmax, Cavg).</li> </ul> |
| Exploratory<br>Analyses | <ul> <li>Change in quantitative influenza viral load over time and change from baseline measured from nasopharyngeal swab samples as determined by qRT-PCR and quantitative virus culture (qVC)</li> <li>Percentage of subjects with no detectable influenza viral RNA by qRT-PCR and qVC.</li> </ul> |
| | Percentage of subjects with co-infected viruses by multiplex RT PCR. |
| | • Percentage by type of co-infected viruses by multiplex RT PCR. |
| | • Quantitative and qualitative changes in exploratory biomarkers (may include but are not limited to: IL-8, procalcitonin, respiratory neutrophil cell counts, neutrophil elastase, and myeloperoxidase). |
| | PK exposure for DNX and pharmacodynamic parameters. |
| | • FLU PRO questionnaire |
| | Activities of daily living (Katz ADL Score) |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Given that the study has been terminated early and only 10 subjects have been enrolled, no formal hypothesis testing will be performed for the study. All analyses will be descriptive and not intended for making definitive conclusions. Only a selected set of originally planned analyses will be performed and all data will be listed.

# 2.2. Study Objective(s) and Endpoint(s)

| | Objectives | Endpoints |
|---|---|---|
| Pri | mary | • |
| • | To assess the efficacy of treatment with IV DNX twice daily given with oral oseltamivir compared to oral oseltamivir twice daily on time to clinical response (TTCR) | Time to Clinical Response (composite) Hospital discharge OR Normalization of: - Temperature; and - Oxygen status; and - Respiratory status/Heart Rate/SBP(normalization of 2 out of these 3 parameters) |
| Sec | condary | |
| • | To assess the efficacy of treatment with IV DNX twice daily given with oral | Time to Respiratory Response defined as meeting at least one criterion below |
| | oseltamivir compared to oral oseltamivir twice daily on time to respiratory response (TTRR) | Return to pre-morbid oxygen requirement (subjects with chronic oxygen use), OR |
| | | Return to no requirement of supplemental oxygen, OR |
| | | Respiratory rate ≤24/min (without supplemental oxygen) |
| • | To evaluate clinical measures of influenza illness following treatment with IV DNX twice daily given with oral oseltamivir compared to oral oseltamivir twice daily | Time to absence of fever |
| | | Time to improved oxygen status |
| | | Time to improved heart rate |
| | | Time to improved SBP |
| | | Proportion of subjects with clinical response over time |
| | | Proportion of subjects with improved respiratory status over time |
| | | Time to improvement of ventilation status: modality, frequencies and durations of invasive and non-invasive ventilator support, duration of oxygen supplementation. |
| | | Length of stay in the ICU |
| | | Frequency of ICU admission and readmission |
| | | Length of stay in the hospital |
| | | Rates of development of septic shock |
| | | Frequency of antibiotic use |

| | Objectives | Endpoints |
|---|---|---|
| | | Proportion of subjects with improvement in Ordinal scale of clinical efficacy over time: Death Mechanical vent In the ICU/ non MV Non-ICU hospitalization Hospital discharge |
| • | To characterize the safety and tolerability of IV DNX twice daily given with oral oseltamivir compared to oral oseltamivir twice daily | Frequency of adverse events (AEs) and serious adverse events (SAEs) Frequency of adverse events of special interest (AESIs) Change from baseline in clinical laboratory |
| • | To characterize the pharmacokinetics of IV DNX in subjects hospitalized for influenza | evaluations, and ECG parameters Standard pharmacokinetic parameters for IV DNX (i.e. AUC, Cmax, Cavg). |
| Ex | ploratory | |
| • | To assess changes in influenza viral load from nasopharyngeal swabs following treatment with IV DNX twice daily given with oral oseltamivir compared to oral OSV twice daily; perform resistance analysis and a multiplex PCR assay with respiratory virus panel to assess coinfection. | Change in quantitative influenza viral load over time and change from baseline measured from nasopharyngeal swab samples as determined by qRT-PCR and quantitative virus culture (qVC) Percentage of subjects with no detectable influenza viral RNA by qRT-PCR and qVC. Percentage of subjects with co-infected viruses by multiplex RT PCR. Percentage by type of co-infected viruses by multiplex RT PCR. Change in quantitative viral load of other virus co-infections over time and change from baseline measured from nasopharyngeal swab samples, as determined by qRT-PCR. Frequency of emergent resistance to OSV |
| • | To explore the effects of IV DNX twice daily given with oral oseltamivir compared to oral OSV twice daily with IV DNX placebo on biomarkers of inflammation and immune response from nasal samples or fluid, endotracheal samples, whole blood, bronchoalveolar lavage, and/or serum. | Quantitative and qualitative changes in exploratory biomarkers (may include but are not limited to: IL-8, procalcitonin, respiratory neutrophil cell counts, neutrophil elastase, and myeloperoxidase). |
| • | To characterize the PK response | PK exposure for DNX and pharmacodynamic |

| Objectives | Endpoints |
|---|---|
| relationship of IV DNX. | parameters. |
| To determine health outcome impact of IV | FLU PRO questionnaire |
| DNX twice daily given with oral OSV compared to oral OSV twice daily | Activities of daily living (Katz ADL Score) |
| compared to oral OSV twice daily | Activity level |
| | Hospital readmission rates |

## 2.3. Study Design

Subjects meeting all eligibility criteria will be randomized 2:2:1 to one of three treatment groups in accordance with the central randomization schedule generated by Clinical Statistics prior to the start of the study, using validated internal software. All randomized subjects will take investigational drug or matching placebo twice daily for up to 5 days in the hospital.

## 2.4. Statistical Hypotheses

No statistical hypotheses will be formally tested.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

An Independent Data Monitoring Committee (IDMC) will perform monitoring and reviews of available safety and efficacy data. Details are specified in the IDMC charter. No formal interim analysis will be performed.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects enrol in the study at the time of study termination have completed the study, which is defined as completing the Day 45 assessment.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to Ramos NG procedures.

## 4. ANALYSIS POPULATIONS

Table 1 Analysis Populations

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Intent to Treat Exposed Population (ITT- E) | Comprised of all randomized subjects who receive at least one dose of investigational product. Subjects will be assessed according to their randomized treatment, regardless of the treatment they receive. | Study Population<br>and disposition |
| Safety | <ul> <li>Comprised of all randomized subjects who receive at least one dose of IP.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | Safety |
| Influenza Positive<br>Population (IPP) | Comprised of all subjects in the ITT-E population with influenza infection (positive influenza PCR or culture at any timepoint) confirmed by central lab testing. | Efficacy, Health Outcomes, Virology, Biomarker |
| PK | Comprised of all subjects who underwent<br>blood PK sampling during the study and from<br>whom one or more blood concentration is<br>determined. | • PK |
| All Subjects<br>Screened | Comprised of all subjects screened for inclusion in the study | Study Population |

#### NOTES:

Please refer to Appendix 13: List of Data Displays which details the population to be used for each display being generated.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Treatment States and Phases |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |
| 11.9 | Appendix 9: Examination of Covariates, Subgroups & Other Strata |
| 11.10 | Appendix 10: Multiple Comparisons & Multiplicity |
| 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 11.12 | Appendix 12: Abbreviations and Trade Marks |
| Error! | Appendix 13: List of Data Displays |
| Referen<br>ce | |
| source | |
| not | |
| found. | |
| 11.14 | Appendix 14: example Mock Shells for Data Displays |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the ITT-E population, unless otherwise specified.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

 Table 3
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data Displays Generate | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition | Υ[1] | | |
| Reasons for Screen Failure | | | Y |
| Reasons for Study Withdrawal | <b>Y</b> [2] | | Υ |
| Reasons for Discontinuation of Study Treatment | Υ | | Υ |
| Subjects for Whom the Treatment Blind was Broken | | | Y |
| Planned and Actual Treatments | | | Υ |
| Protocol Deviations | | | |
| Important Protocol Deviations | | | Υ |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Y [3] |
| Populations Analysed | | | |
| Study Populations | Υ | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | <b>Y</b> [1] | | Υ |
| Race and Racial Combinations | Υ | | <b>Y</b> [4] |
| Prior and Concomitant Medications | | | |
| Concomitant Medications | | | Υ |
| Prior Exposure to Oseltamivir | | | Υ |
| Exposure | | | |
| Exposure to Study Treatment | Υ | | Υ |
| Other | | | |
| Flu Details (includes influenza subtypes) | <b>Y</b> [1] | | Υ |
| Past and Current Medical Conditions | Υ | | Υ |
| Chronic underlying illness at baseline for Subjects with Renal Impairment | | | <b>Y</b> [5] |
| Ventilation and Oxygenation Status at Baseline and Any Time | Y | | Y |
| Chest X-ray at Baseline | | | Υ |


201023

| Endpoint / Parameter / Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Table Figure |

## NOTES:

- Y = Yes display generated.
  [1] For ITT-E and IPP
  [2] Included in the Summary of Subject Disposition
  [3] Listing also includes analysis population exclusions.
  [4] Listing of race
  [5] Panel impointment
- [5] Renal impairment is based on Creatinine Clearance Criteria .

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Efficacy Analyses

The primary efficacy analyses will be based on the IPP population, unless otherwise specified. Table 5 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

## 7.1.1. Overview of Planned Efficacy Analyses

Table 4 Overview of Planned Primary Efficacy Analyses

| Endpoint | Stats Analysis | | | Summary | | Indiv | idual |
|---|---|---|---|---|---|---|---|
| 1 | Т | F | L | Т | F | F | L |
| | Absolute | | | | | | |
| Time to Clinical Response (TTCR) | | | | <b>Y</b> [1] | | | Υ |
| Proportion of Subjects Achieving Improved Clinical | | | | <b>Y</b> [1] | | | |
| Response by End of Study | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- [1]. Proportion of clinical response and Kaplan Meier estimates for the median of TTCR for each treatment group and 95% CI will be provided

## 7.1.2. Planned Efficacy Statistical Analyses

The clinical response is defined as hospital discharge due to clinical improvement or meeting following vital signs/ventilation criteria.

| Sign of clinical response | Response criteria |
|---|---|
| Temperature <sup>1</sup> | ≤36.6°C (≤97.9°F) – axilla/temporal, or |
| | ≤37.2°C (≤99°F) – oral, or |
| | ≤37.7°C (≤99.9°F) – rectal/core <sup>5</sup> , tympanic |
| AND | |
| Oxygen saturation <sup>2,3</sup> | ≥95% (without supplemental oxygen) |
| AND 2 out of the following | ng 3 criteria: |
| Respiratory status | For subjects with chronic hypoxia and supplemental oxygen use: return to pre-morbid oxygen requirement, OR |
| | For subject with supplemental oxygen use at study entry: need for supplemental oxygen (administered by any modality – ventilator, non-invasive ventilation, facemask, face-tent, nasal canula, etc) to no need for supplemental oxygen, OR |
| | • For subject without supplemental oxygen use and respiratory rate > 24/min at study entry: respiratory rate ≤24/min |
| Heart rate | ≤100/min |
| Systolic blood pressure <sup>4</sup> | ≥90 mmHg |

- 1. Without the use of antipyretics within 8 hours
- 2. A subject with a history of chronic hypoxia (without supplemental oxygen) will satisfy normalization criteria for oxygen saturation if the value (without supplemental oxygen) is ≤2% from subject's historical oxygen saturation baseline as recorded within 12 months prior to enrolment as documented in the subject's medical records.
- 3. This requirement will be waived for subjects with a history of chronic supplemental oxygen requirement who have a baseline oxygen saturation <95% with supplemental oxygen, within 12 months prior to enrolment as documented in the subject's medical records.
- 4. Without inotropic support administered within 2 hours.
- 5. Core temperatures include rectal, indwelling catheters and Swan Ganz catheters.

## **Statistical Analyses**

#### Endpoint(s)

• Time to Clinical Response (TTCR), days.

#### **Derivation of TTCR**

The clinical response based on vital signs/ventilation status requires 24-hour confirmation. Considering 2-hour assessment window, the response confirmation period is 22 hours, i.e. all assessments within 22 hours of the initial response and at least one at or beyond 22 hours need to meet the criteria in order for the response to be confirmed. Any missing scheduled assessment will be imputed with response value of 0 (1 means response). Only hospital discharge due to clinical response or a confirmed response based on vital signs/ventilation criteria is considered as event for the TTCR analysis. Hospital discharge due to clinical improvement can serve as 24-hour confirmation for the clinical response and the event date should be the onset of the vital signs response. Subjects who died prior to achieving a clinical response will be assigned a worst value of TTCR (99 days). All other subjects who did not achieve a confirmed response will be censored at the last assessment date of vital signs.

For further details of the calculation of TTCR see Section 11.6.4.

### **Model Specification**

Not applicable

## **Model Checking & Diagnostics**

Not applicable

#### **Model Results Presentation**

Not applicable

### **Sensitivity and Supportive Statistical Analyses**

 No sensitivity analyses or subgroup analyses will be performed given the small number of subjects.

### 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Efficacy Analyses

## 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the IPP population, unless otherwise specified. Table 5 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 13: List of Data Displays. Given the small number of subjects, only time to respiratory response will be summarized. Data relevant to other secondary endpoints will be listed including vital signs, ventilation status, hospital discharge, hospital re-admission, and ICU stay.

Table 5 Overview of Planned Secondary Efficacy Analyses

| Endpoint | Stats Analysis | | | Analysis Summary | | ummary Individua | |
|---|---|---|---|---|---|---|---|
| | Т | F | L | T | F | F | L |
| | Absolute | | | | | | |
| Time to Respiratory Response (TTRR) | | | | <b>Y</b> [1] | | | |

<sup>[1]</sup> Proportion of clinical response and Kaplan Meier estimates for the median of TTCR for each treatment group and the median difference and 95% CI between two comparisons: each DNX arm and OSV will be provided

## 8.2. Safety Analyses

## 8.2.1. Overview of Planned Adverse Events Analyses

The safety analyses will be based on the Safety population, unless otherwise specified. The summaries include on-treatment and post-treatment assessments unless otherwise noted.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 6 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Absol | ute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and Maximum Grade | Υ | | Υ |
| All AEs by Overall Frequency | Υ | | |
| Grade 2-4 AEs by Overall Frequency | Υ | | |
| All Drug-Related AEs by Overall Frequency | Υ | | |
| All Non-Serious AEs by Overall Frequency | Υ | | |
| Drug-Related Grade 2-4 AEs by Overall Frequency | Υ | | |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Y |
| Listing of Adverse Events for Subjects with Neutropenia by Grade (>=Grade 1) | <b>Y</b> [1] | | |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs | | | Y |
| Non-Fatal Serious AEs | Υ | | Υ |
| Serious AEs by SOC | Υ | | |
| Reasons for Considering as a Serious AE | | | Y |
| Drug-Related Non-Fatal Serious AEs | Υ | | |
| Drug-Related Serious AEs by SOC | Υ | | |
| Adverse Events Leading to Withdrawal from Study by Overall Frequency | | | Υ |
| Adverse Events Leading to Permanent Discontinuation of Study Treatment by | | | Υ |
| Overall Frequency | | | 1 |
| Summary of Serious Adverse Events by System Organ Class and Preferred | Υ | | |

| Endpoint / Parameter/ Display Type | Absolute | | ute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Term (Number of Subjects and Occurrences) | | | |
| Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Y | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]. Toxicity Grading is based on the Division of AIDS Grading (Section 12.5 of the protocol)

## 8.2.2. Overview of Planned Clinical Laboratory Analyses

The safety analyses will be based on the Safety population, unless otherwise specified. The summaries include on-treatment and post-treatment assessments unless otherwise noted.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 7 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Absolute | | | ange | from BL |
|---|---|---|---|---|---|---|
| | Sum | Summary Individ | | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Summary of Data Supporting Safety Halting Criteria | <b>Y</b> [1] | | | | | |
| Chemistry Changes from Baseline | | | | Υ | | |
| Creatinine by Visit | Υ | Υ | | Υ | | |
| Hematology Changes from Baseline | | | | Υ | | |
| Individual Plot of Absolute Neutrophils Count by Visit by Subject | | Υ | | | | |
| All Laboratory | _ | | | | | |
| Summary of Maximum Treatment Emergent Toxicities of All Lab Parameters | Υ | | | | | |
| Laboratory Data Abnormalities of Potential Clinical Importance (Grade 3-4) | | | | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- [1] Summary includes the proportion of subjects with creatinine increase of 0.5 mg/dl on 2 consecutive visits

## 8.2.3. Overview of Planned Other Safety Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 8 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abso | olute | Change from B | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Summary | | Summary | | Individual | Sumr | nary | Individual |
| | Т | F | L | T F | | L | | | | |
| ECG | | | | | | | | | | |
| All ECG Values for Subjects with a Value of PCI <sup>[1]</sup> | | | Y | | | | | | | |
| Abnormal ECG Findings[2] | | | Y | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] When QTc data is evaluated for PCI, all of the QTcB, QTcF and QTc collected in the eCFR are considered. Any one of the three meeting the PCI range is identified as an ECG event of PCI..
- [2] When QTc data is evaluated for ECG abnormality, all of the QTcB, QTcF and QTc collected in the eCFR are considered. Any one of the three meeting the abnormality criteria is identified as an abnormal ECG Finding.

## 8.3. Pharmacokinetic Analyses

## 8.3.1. Overview of Planned Pharmacokinetic Analyses

PK samples will be drawn on Day 1 (pre-dose, prior to 2<sup>nd</sup> dose), Days 3 and 5 to coincide with PD measurements (biomarkers) and additionally drawn on Day 3 (5<sup>th</sup> or 6<sup>th</sup> dose) at 0.5, 1 (end of infusion), 1.5, 2, 3, 4, 8 and 12 hours post-dose.

Table 9 provides an overview of the planned analyses with full details being presented in Appendix 13: List of Data Displays.

Table 9 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untransformed | | | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | T | F | L | F | T | F | L |
| DNX Concentrations | Υ | Υ | | Υ | Υ | Y | | |
| DNX PK Parameters | | Υ | | Υ | | Y | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.3.2. Drug Concentration Measures

Concentrations of Danirixin (GSK1325756) in blood will be listed and summarised by treatment group, day and nominal time.

Individual blood concentration-time profiles and median/mean profiles by treatment group will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Process & Standards).

### 8.3.3. Pharmacokinetic Parameters

### 8.3.3.1. Deriving Pharmacokinetic Parameters

Pharmacokinetic parameters described in Table 10 will be determined from the concentration-time data, as data permits.

Table 10 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-12) | Area under the concentration-time curve from time zero to the time of the |
| | last quantifiable concentration (C(t)) will be calculated using the linear |

| Parameter | Parameter Description |
|---|---|
| | trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Cavg | Average concentration. |

## 8.3.3.2. Statistical Analysis of Pharmacokinetic Parameters

No formal statistical analysis of derived pharmacokinetics parameter will be performed.

## 8.3.4. Population Pharmacokinetic (PopPK) Analyses

Given the small number of subjects enrolled population PK analysis for this study will not be performed.

## 8.4. Biomarker Analyses

## 8.4.1. Overview of Planned Biomarker Analyses

The Biomarker analyses will be based on the Influenza Positive Population, unless otherwise specified.

Table 11 provides an overview of the planned Biomarker analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 11 Overview of Planned Biomarker Analyses

| [Endpoint / | Untransformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | Abso | olute | | ( | Change fro | m Baselin | ie |
| Type] | Summary | | Indiv | Individual | | mary | Individual | |
| | T | F | F | L | T | F | F | L |
| Serum Biomarkers | | | Υ | Υ | | | | |
| Nasal wash<br>biomarkers <sup>[1]</sup> | | | Y | Y | | | | |
| Nasal SAM strips biomarkers | | | Y | Y | | | | |
| BAL Biomarker | | | Υ | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

[1] includes neutrophil count

## 8.5. Pharmacodynamic / Biomarker Statistical Analyses

## 8.5.1. Overview of Planned Pharmacodynamic / Biomarker Analyses

The Pharmacodynamic / Biomarker analyses will be based on the Influenza Positive Population, unless otherwise specified.

Table 12 provides an overview of the planned Biomarker / Pharmacodynamic analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 12 Overview of Planned Pharmacodynamic / Biomarker Analyses

| | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Individual | | Summary | | Individual | |
| | Η | F | F | Ш | Т | F | F | L |
| Biomarkers vs. Biomarkers | | | <b>Y</b> [1] | | | | | |
| Area under the curve for Serum Biomarkers TTCR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for Nasal wash biomarkers – TTCR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for Nasal SAM Strips biomarkers – TTCR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for BAL biomarkers – TTCR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for Serum Biomarkers - TTRR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for Nasal wash biomarkers – TTRR | | | <b>Y</b> [2] | | | | | |
| Area under the curve for Nasal SAM biomarkers – TTRR | | | <b>Y</b> [2] | | _ | | | |
| Area under the curve for BAL biomarkers – TTRR | _ | | <b>Y</b> [2] | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Matrix comparative plot of individual scatter plot of biomarkers vs. biomarkers for Each Biomarker. The x and the y-axis will include Serum, Nasal Wash, Nasal SAM Strips and BAL. Include the Pearson's correlation coefficient and p-value.
- [2] Individual scatter plot of area under the curve biomarkers vs Time to Clinical Response, Time to Respiratory Response.

## 8.6. Pharmacokinetic / Pharmacodynamic Analyses

Relationships between Danirixin systemic exposure and the following pharmacodynamic measures will be explored graphically:

• Target engagement biomarker: IL-8, respiratory neutrophil cell counts, neutrophil elastase, and myeloperoxidase.

Pharmacokinetic/pharmacodynamic modelling may be attempted to describe any relationship including appropriate models for longitudinal variables versus systemic exposure. Results of PK/PD modelling analysis will be done under a separate Reporting and Analysis Plan and will be reported separately from the main CSR.

## 8.7. Health Outcome Analyses

## 8.7.1. Overview of Planned Health Outcome Analyses

The health outcome analyses will be based on the IPP population, unless otherwise specified.

 Table 13
 Overview of Planned Health Outcome Analyses

| Endpoints | Absolute | | | | Change from BL | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | T | F | L | F | Τ | F | L |
| KATZ ADL | | | | Y | | Y | | |
| Flu PRO | | Υ | | Υ | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 9. VIROLOGY ANALYSES

# 9.1. Overview of Planned Virology Analyses

The virology analyses will be based on the IPP population, unless otherwise specified.

Table 14 provides an overview of the planned analyses, with full details being presented in Appendix 13: List of Data Displays.

Table 14 Overview of Planned Virology Analyses

| Endpoints | Absolute Change from BL | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | Т | F | L | F | T | F | L |
| Influenza Viral Load by qRT-<br>PCR | | | | Y | | <b>Y</b> [2,3] | Υ[1,2,3] | |
| Influenza Viral Load by qVC | | | | Υ | | <b>Y</b> [2,4] | <b>Y</b> [1,2,4] | |

| Endpoints | | Abs | olute | | Change from BL | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | Т | F | L | F | Т | F | L |
| Resistance Associated Mutations Detected in the NA Gene by Subtype Nasopharyngeal | | Υ | | Y | | | | |
| Resistance Associated Mutations Detected in the HA Gene by Subtype Nasopharyngeal | | Y | | Y | | | | |
| Proportion of Subjects - Positive Other Viruses by Multiplex | | Y | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Change from baseline plot for nasopharyngeal
- [2] For nasopharyngeal
- [3] Overall virus and by subtype
- [4] For subjects culture positive at baseline, if warranted.

# 9.2. Planned Virology Statistical Analyses

qVC data will be summarized for subjects who are culture positive at baseline. For the RT-PCR summaries for Flu A and Flu B combined, coinfected subjects values will be averaged.

The following is a list of viruses detected in the multiplex assay:

- Adenovirus
- Coronavirus 229E
- Coronavirus HKU1
- Coronavirus OC43
- Coronavirus NL63
- Human Metapneumovirus
- Human Rhinovirus/Enterovirus
- Influenza A
- Influenza A/H1
- Influenza A/H1-2009
- Influenza A/H3
- Influenza B
- Parainfluenza 1

- Parainfluenza 2
- Parainfluenza 3
- Parainfluenza 4
- RSV A+B

For the viruses with multiple subtypes, the data will be summarized by same virus family (e.g. corona virus, parainfluenza, and RSV, influenza A)

The list of mutations which includes but is not limited to H275Y will be provided only if the data is available.

# 10. REFERENCES

FDA. *Guidance for Industry*. Center for Drug Evaluation and Research, United States Food and Drug Administration; 1999. Population Pharmackinetics.

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Assessment Windows |
| Section 11.4 | Appendix 4: Treatment States & Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | <ul> <li>Baseline Definitions &amp; Derivations</li> </ul> |
| | Reporting Process & Standards |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | • Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 11.9 | Appendix 9: Examination of Covariates and Subgroups |
| Section 11.10 | Appendix 10: Multiple Comparisons and Multiplicity |
| Section 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 11.13 | Appendix 13: List of Data Displays |
| Section 11.14 | Appendix 14: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

No Per Protocol Population will be used in the analysis.

# 11.2. Appendix 2: Time & Events

### 11.2.1. Protocol Defined Time & Events

Table 15 Time and Events Table: Assessments at Baseline and During Treatment

| | Eligibilit<br>y<br>Assess<br>ments | | During Treatment - 5 days <sup>a</sup><br>Inpatient | | | | | |
|---|---|---|---|---|---|---|---|---|
| Procedures | | Baselin<br>e/<br>Study<br>Day 1ª | Study<br>Day 2 | Study<br>Day 3 | Study Day 4 | Study Day<br>5 /day of<br>last dose <sup>a</sup> | Study<br>Day 6 if<br>applicab<br>le <sup>b</sup> | |
| Written informed consent | Х | X | | | | | | |
| Subject demography | Х | X | | | | | | |
| Physical examination <sup>c</sup> | | X | Х | Х | Х | Х | Х | Daily |
| Influenza Test – locally performed (equipment provided by GSK) | Х | X | | | | | | |
| Medical/Prior<br>Medication/Drug/Smoking<br>History | Х | X | | | | | | |
| HIV and Liver Disease<br>History <sup>d</sup> | Х | Х | | | | | | |
| Influenza symptomse | X | X | | | | | | |
| HIV, Hep B and Hep C<br>Test <sup>f</sup> | Х | | | | | | | |
| Chronic underlying illness assessment | X | Х | | | | | | |
| Inclusion/Exclusion Criteria | Х | | | | | | | |
| Safety/Efficacy<br>Assessments | | | | | | | | |
| Chest X-ray <sup>g</sup> | | X | | | | | | |
| ECG <sup>h</sup> | Х | X | | | | Х | Х | |
| Adverse events | | X | X | X | X | Х | Х | Daily |
| Concomitant medications <sup>i</sup> | | X | Х | Х | X | X | Х | Daily |
| Complications of influenza/associated antibiotic use <sup>j</sup> | | X | Х | X | Х | X | Х | Daily |
| Vital signs<br>(temperature, HR, BP,<br>respiratory rate,<br>oxygen saturation,<br>ventilation status) <sup>k</sup> | Х | Х | Х | Х | X | Х | Х | 3 x Daily |

| | Eligibilit<br>y<br>Assess<br>ments | | During Treatment - 5 days <sup>a</sup><br>Inpatient | | | | | |
|---|---|---|---|---|---|---|---|---|
| Procedures | | Baselin<br>e/<br>Study<br>Day 1ª | Study<br>Day 2 | Study<br>Day 3 | Study Day 4 | Study Day<br>5 /day of<br>last dose <sup>a</sup> | Study<br>Day 6 if<br>applicab<br>le <sup>b</sup> | |
| Flu PRO | | X | X | X | X | X | Х | Daily |
| Katz Activities of Daily Living | | Х | Х | Х | Х | Х | Х | Daily |
| Activity level <sup>m</sup> | | Х | Х | Х | Х | Х | Х | Daily |
| Chemistry including Liver Function Tests (Local+Central) <sup>n</sup> | X | Х | | Х | | X | Х | Day 6,7,8 |
| Serum creatinine<br>(Local+Central) ° | Х | Х | Х | Х | Х | Χ | Х | Day<br>6,7,8 |
| Hematology<br>(Local+Central) p | Х | Х | | Х | | Х | Х | Day 6,7,8 |
| Urine Output q | | Х | Х | Х | χ | Х | Х | |
| Pregnancy testr | Х | Х | | | | | | PT Day<br>3 |
| Nasopharyngeal swabs | | X | | Х | | X | X | Day<br>8,12,16,<br>20,24,28<br>,32 |
| Nasal Swab <sup>t</sup> | Х | X | | | | | | |
| BAL <sup>u</sup> | | X | | X | | X<br>X | X | |
| Endotracheal aspirate <sup>v</sup> | | Х | | X | | X | X | Day<br>8,16,24,<br>32, 45 |
| Nasal SAM strips<br>(biomarkers) <sup>w</sup> | | X | | Х | | X | X | Day<br>8,16,24,<br>32,<br>dischar<br>ge or<br>Day 45 |
| Nasal washes <sup>x</sup> | | Х | | Х | | Х | Х | Day<br>8,16,24,<br>32,<br>dischar<br>ge or<br>Day 45 |
| Exploratory Biomarkers (Blood Sample) | | X | | Х | | X | Х | Day<br>8,16,24,<br>32,<br>dischar<br>ge or<br>Day 45 |
| PK sample (Dried Blood Spot) <sup>y</sup> | | Х | | Х | | X | X | |
| Genetics Sample (Blood Sample) <sup>z</sup> | | Х | | | | | | |
| Transcriptomics (Blood Sample) <sup>z</sup> | | X | | Х | | X | Х | Day 8,<br>16, 24, |

| | Eligibilit<br>y<br>Assess<br>ments | | During Treatment - 5 days <sup>a</sup><br>Inpatient | | | | | |
|---|---|---|---|---|---|---|---|---|
| Procedures | | Baselin<br>e/<br>Study<br>Day 1 <sup>a</sup> | Study<br>Day 2 | Study<br>Day 3 | Study Day 4 | Study Day<br>5 /day of<br>last dose <sup>a</sup> | Study<br>Day 6 if<br>applicab<br>Ie <sup>b</sup> | |
| | | | | | | | | 32,<br>dischar<br>ge or<br>Day 45 |
| Study Treatments | | | | | | | | |
| Administration of investigational medication (IV) and oseltamivir (oral) twice daily | | X | X | X | X | X | X | |

- a. A 'Day' is defined as a 24 hour period (Treatment Day), therefore depending on the start time of the first dose of IV DNX, a Treatment Day may span two calendar days.
- Day 6 assessments only applicable if last day of dose of randomized treatment is on Day 6 (i.e for subjects who
  received first dose after 12 noon on Baseline/Day 1.
- c. Physical exam to be performed twice daily for subjects in the sentine cohort.
- d. Enrollment into the study will be based on history of diagnosis of HIV and liver disease. Blood samples will be analyzed after enrollment to retrospectively determine if subject is HIV, Hep B or Hep C postivie; however, results will not be available until after completion of dosing.
- e. Influenza symptoms to be assessed only at baseline for inclusion.
- f. Enrollment into the study will be based on any history of diagnosis of HIV and liver disease.
- g. Chest X-ray at Baseline and whenever clinically indicated.
- h. ECG: For the ECG on Baseline/Day 1, one 12-lead ECG (can be done within approximately 24 hours prior to dosing). At Baseline and on Day 5 or last treatment day, a monitoring strip can be utilized if a 12-lead ECG cannot be performed.
- i. Concomitant medications for influenza treatment of the current episode to be recorded from Day -7 (i.e. one week prior to baseline), if available.
- Complications of influenza such as bacterial pneumonia, pneumothorax, pleural effusion, ARDS, myositis, encephalitis, myocarditis, and associated antibiotic use will be recorded on all assessment days.
- k. Vital signs and ventilation status to be assessed three times daily during the treatment period between approximately 8 AM and 8 PM.
- I. Katz ADL score collected once daily while hospitalized.
- M. Activity level to be recorded as one of three responses (bed rest, limited ambulation or unrestricted) everyday while hospitalized
- n. Chemistry panel including Liver Function Tests to be required once every other day during treatment (local testing (L) of LFTs for subject management as well as central laboratory testing (C)).
- Serum creatinine level required at Baseline and twice daily during treatment for subjects in the sentinel cohort. For all other subjects, serum creatinine level required at Baseline and once daily during treatment (local testing (L) for subject management as well as central testing(C)).
- Hematology panel including CBC with differential required every other day during treatment (local testing (L) for subject management as well as central testing(C))
- q. Urine output to be measured twice daily for subjects in the sentinel cohort.
- r. Ultrasensitive urine or blood pregnancy test required in women of childbearing potential prior to dosing and 3 days post last dose of study treatment.
- s. Nasopharyngeal swab will be used for influenza Subtype RT-PCR, qRT-PCR, quantitative culture and may also be used for rapid influenza diagnosis; Will also be used for viral genotyping and phenotyping if needed and multiplex PCR assay.
- t. Nasal swab collected for influenza diagnostic test or other local test for influenza diagnosis

- BAL samples (for biomarkers) are requested only if the procedure/sampling is being carried out for routine
  management of the patient and at any timepoint throughout the study
- Endotracheal aspirates (biomarkers/neutrophil counts) are required for subjects who are intubated.
- w. Nasal samples for biomarkers will be collected at the days indicated from all subjects using nasal SAM strips.
- x. An optional procedure, nasal wash, will be used to collect nasal samples from as many non-intubated subjects as feasible.
- y. PK samples will be drawn on Day 1 (pre-dose), Days 3 and 5 to coincide with PD measurements (nasal washes if done, endotracheal samples and a blood draw for exploratory biomarkers). In sentinel cohort 1 (less severe subjects with normal renal function), PK samples will be additionally drawn on Day 3 at pre-dose, and 0.5, 1 (end of infusion), 1.5, 2, 3, 4, 8 and 12 hours post-dose. **Note: PK draws must be collected from the opposite arm from the infusion arm.**
- z. Informed consent for optional substudies (e.g., genetic research and transcriptomics), must be obtained before collecting samples. In subjects who consent, a blood sample for genetic research is collected at the baseline visit, or at the earliest point possible during the treatment period for genetic research testing; blood samples for transcriptomics are taken on each of the indicated days and used to evaluate changes in transcriptome profiles.

Table 16 Time and Events Table: Post-Treatment and Post-Discharge Assessments

| | Post-Discharge Visits/TCs and Assessments Outpatient a | | | | | |
|---|---|---|---|---|---|---|
| Procedures | PT Day 3<br>(Visit) | Study<br>Day 8<br>(TC) | Study<br>Day<br>15<br>(TC) | Study Day 22<br>(TC) | Study Day<br>30 (TC) | Study Day 45<br>(Visit) |
| Safety/Efficacy<br>Assessments | | | | | | |
| Adverse events | Х | Χ | Х | Х | Х | Х |
| Concomitant medications | Х | Χ | Х | Х | Х | Х |
| Brief Physical Exam | Х | | | | | X |
| Complications of influenza / associated antibiotic use <sup>b</sup> | Х | X | Х | Х | Х | X |
| Temperature | Х | Х | Х | Х | Х | Х |
| Other Vital signs (HR, BP, respiratory rate, oxygen saturation, ventilation status) <sup>c</sup> | Х | | | | | Х |
| Flu PROd | Daily<br>through Day<br>14 | Daily<br>through<br>Day 14 | Х | Х | Х | Х |
| Katz Activities of Daily Livinge | Х | X | Х | X<br>X | Х | X |
| Activity level <sup>f</sup> | Daily<br>through Day<br>14 | Daily<br>through<br>Day 14 | X | Х | Х | Х |
| Laboratory Assessments | | | | | | |
| Clinical chemistryincluding LFTs <sup>9</sup> (Local+Central) | X | | | | | X |
| Serum Creatinineh<br>(Local+Central) | Х | | | | | Х |
| Hematology <sup>i</sup><br>(Local+Central) | Х | | | | | Х |
| Pregnancy testi | Х | | | | | |
| Nasopharyngeal swabs | Х | | | | | |
| Exploratory Biomarkers (Blood Sample) <sup>k</sup> | Х | | | | | Х |
| Transcriptomics (blood | Х | | | | | X |

| sample) <sup>I</sup> | | | | | | |
|-----------------------------|---|---|---|---|---|---|
| Nasal SAM strips | Х | | | | | Х |
| (biomarkers) <sup>m</sup> | | | | | | |
| Nasal washes <sup>m</sup> | Х | | | | | Χ |
| Hospital Readmission Status | Х | Χ | Х | Х | Х | X |

- a. Following discharge from hospital, outpatient clinic visit/TC schedule of assessments will be followed for those patients who are discharged before Day 45. For 5 days treatment, PT Day 3 will be the same as Day 8 and will be a clinic visit.
- b. Complications of influenza such as bacterial pneumonia, pneumothorax, pleural effusion, ARDS, myositis, encephalitis, myocarditis, and associated antibiotic use will be recorded on all assessment days.
- c. Vital signs and ventilation status will be assessed at clinic visits (PT Day 3 and Day 45).
- d. FLU PRO to be measured once daily through Study Day 14.
- e. Activities of Daily Living (Katz Scale) to be done at clinic visits and at TCs.
- f. Activity level assessed by reporting on a 3 point scale of bed rest (1), limited ambulation (2) or unrestricted (3) to be done daily through Study Day 14.
- g. Clinical chemistry including LFTs to be required once every other day until PT Day 3 (for LFTs, local testing for subject management until PT Day 3; central testing for all assessments, including at Day 45).
- h. Serum creatinine required once every day until PT Day 3 (local testing for subject management until PT Day 3; central testing for all assessments, including at Day 45).
- i. Hematology panel including CBC with differential required once every other day until PT Day 3 (local testing for subject management until PT Day 3; central testing for all assessments, including at Day 45).
- j. Ultrasensitive urine pregnancy test required in women of childbearing potential on PT Day 3.
- k. Blood samples will be collected for exploratory biomarkers at PT Day 3, and at Study Day 45.
- I. Blood samples for transcriptomics will be collected on PT Day 3 and Study Day 45 and are optional. Samples will be collected only from those subjects who provide informed consent for genetic research.
- m. Nasal samples for biomarkers will be collected at PT Day 3 and Study Day 45 from all subjects using nasal SAM strips. In addition, an optional procedure, nasal wash, will be used to collect nasal samples from as many non-intubated subjects as feasible.

# 11.3. Appendix 3: Assessment Windows

This study will not use assessment windows.

# 11.4. Appendix 4: Treatment States and Phases

#### 11.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date< Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### 11.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

### 11.4.2.1. Treatment States for Concomitant Medications Data

| Treatment State | Definition |
|---|---|
| Pre- Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post Treatment | Date > Study Treatment Stop Date |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment. "On-Study" is considered assessment on-treatment and post-treatment.

#### 11.4.2.2. Treatment States for AE Data

Unless otherwise noted, AE summaries will include both On-Treatment and Post-Treatment AEs.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date [+ Lag Time] |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Drug-related | If relationship is marked 'YES' on InForm OR value is missing |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

## 11.5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| <u>A</u> | 15 mg FBE IV DNX BID +75 mg OSV<br>BID | 15 mg DNX +OSV | 2 |
| <u>B</u> | 50 mg FBE IV DNX BID + 75 mg OSV<br>BID | 50 mg DNX +OSV | 3 |
| <u>C</u> | IV DNX placebo BID + 75 mg OSV<br>BID | PBO + OSV | 1 |

### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

#### 11.5.2. Baseline Definition & Derivations

#### 11.5.2.1. Baseline Definitions

| Parameter | | nts Considered As<br>eline | Baseline Used in Data |
|---|---|---|---|
| | Screening | Day 1 | Display |
| Vital Signs (temperature, HR, BP, respiratory rate, oxygen status, ventilation status) | Х | Х | Day 1 |
| 12 Lead ECG | Х | Х | Day 1 |
| Laboratory parameters | Х | X | Day 1 |
| Nasopharyngeal Swab | | X | Day 1 |
| Nasal Swab | Х | X | Day 1 |
| Nasal SAM strips (biomarkers) | | X | Day 1 |
| Nasal wash biomarker | | X | Day 1 |
| BAL biomarkers | | Х | Day 1 |
| Serum Biomarkers | | X | Day 1 |
| Katz ADL | | X | Day 1 |
| Flu PRO | | X | Day 1 |

For all endpoints (unless stated otherwise) the baseline value will be the latest pre-dose assessment. This is generally expected to be from the Day 1 visit, although such values may be missing or unscheduled assessments may be performed before treatment start.

## 11.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

## 11.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | Software |
| The currently support to the currently su | The currently supported versions of SAS and TSCG software will be used. |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Area | : \ARPROD\GSK1325756\MID201023\Final_xx |
| QC Spreadsheet : \ARWORK\GSK1325756\MID201023\Final_xx\documents | |
| Analysis Datasets | |

#### **Reporting Process**

- Final analysis and IDMC datasets will be created based on Integrated Data Standards Library (IDSL).
- RTF files will be generated for final analysis.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
  - Unscheduled visits will be included in the maximum toxicity or maximum change from baseline for toxicity tables.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) |

| Reporting Standards | |
|---|---|
| Summary Statistics | of logged data and between geometric coefficient of variation (CVb (%)) will |
| (Log Transformed) | be reported. |
| | ○ $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of log transformed data) |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13 | |

# 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a visit the value closest to the planned/target day for that visit will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Treatment Start Date**

Treatment start date is defined as follows:

 Treatment start date is the date entered onto the IP exposure CRF for when study treatment started.

### Study Day

- Calculated as the number of days from initial study treatment start date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) + 1

Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Post-baseline

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.

# 11.6.2. Study Population

### **Demographics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date.
- Birth date will be presented in listings as 'YYYY'.
#### **Demographics**

Completely missing dates of birth will remain as missing, with no imputation applied.
 Consequently, the age of the subject will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

If not already provided, BMI will be calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 11.6.3. Safety

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- Machine-read values of RR, QTcB or QTcF should not be replaced with re-derived values
- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- Influenza Virus load data from Viroclinics will be imputed as following:
- LLOQ and LLOD per subtype are dependent on the data, assume the values are x.xx,
   y.yy, z.zz, and w.ww for LLOQ, LLOD for qPCR A and q PCR B, respectively

#### **ECG Parameters**

- qPCR A: LLOQ=: x.xx log vp/ml, LLOD: y.yy log vp/ml
  - When CT neg (i.e. qPCRA<LLOD), impute y.yy 0.01</li>
  - When qPCRA between LLOD and LLOQ, impute x.xx 0.01
  - When qualitative results are derived from qPCR: when CT is positive value then "Virus detected" and when CT is neg then "Virus not detected".
- qPCR B: LLOQ: z.zz log vp/ml, LLOD:w.ww log vp/ml
  - When CT neg (i.e. qPCRB <LLOD), impute w.ww 0.01.
  - When qPCRB between LLOD and LLOQ, impute z.zz 0.01
  - When qualitative results are derived from qPCR: when CT is positive value then "Virus detected" and when CT is neg then "Virus not detected".
- TCID50: LLOQ = 0.75
  - $\circ$  When <0.75 impute 0.75 0.01 = 0.74.
  - When qualitative results are derived from <u>TCID50</u>: when TCID50 <0.75 impute "No Virus Isolated", when >0.75 impute "Virus Isolated".
- For other laboratory values, if laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

## 11.6.4. Efficacy

#### **Time to Clinical Response (TTCR)**

TTCR will be derived as detailed in Section 7.1.2 The following is further considerations for the derivation of TTCR

- If an assessment time is missing the following times will be used in the calculation of TTCR: 8:00, 14:00, 20:00 respectively for morning, afternoon and evening assessments. The imputation will not be done for the study day 1.
- If the subject was discharged but is missing the date of discharge then the latest day from individual components will be used. If subject was discharged but the time of discharge is missing, 12:00 time will be used.
- If the subject withdraws consent on the same day as hospital discharge, TTCR will not be considered a failure.

- Deaths which occur after clinical response will not be considered a failure
- When a subject met vital sign criteria and was discharged from hospital during the 24 hour period of stability confirmation, the time of achieving TTCR was defined as the initial time at which vital signs were resolved and not the time of hospital discharge.
- If the clinical response has not been achieved by study completion, TTCR will be censored at the last assessment date of vital signs.
- If the subject did not achieve a clinical response the reason for censoring will be summarized (i.e. did not achieve vital sign resolution or reason for prematurely discontinuing the study).

### Time to Respiratory Response (TTRR)

- Time to Respiratory Response defined as the first time meeting below, for at least 24 hours:
  - o Return to pre-morbid oxygen requirement (subjects with chronic oxygen use), OR
  - Need for supplemental oxygen (administered by any modality ventilator, noninvasive ventilation, facemask, facetent, nasal canula, etc) to no need for supplemental oxygen, OR
  - Respiratory rate >24/min and no supplement oxygen at baseline, and post baseline respiratory rate ≤24/min (without supplemental oxygen)
- Subjects who meet the above criteria at baseline (i.e., normal respiratory response) will not be included in the Kaplan Meier analysis and these subject not be considered as "improved" in the response rate
- If the symptoms have not resolved at Day 45, it will be censored at Day 45.

#### 11.6.5. Biomarker

#### 11.6.5.1. Biomarkers and Source

| SAM | Serum | Nasal Wash | BAL |
|---|---|---|---|
| IL-6, IL-10, IP-<br>10, IL-8, MPO,<br>NE, IL-1b | Procalcitonin | IL-6, IL-10, <b>IP-10</b> , <b>IL-8</b> , <b>MPO</b> , <b>NE</b> , IL-1b | IL-6, IL-10, <b>IP- 10</b> , <b>IL-8</b> , <b>MPO</b> , <b>NE</b> , IL- 1b |
| | C1M, C3M, EL-NE | Neutrophil Cell<br>Counts | |
| SP-D, sRAGE, | SP-D, sRAGE | SP-D, sRAGE | SP-D, sRAGE |

#### Biomarker

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</p>

#### **AUC of Biomarker**

- The area under the curve (AUC) to Day 5, Day 45, and PT Day 3 of biomarker as measured by the level of biomarker from biomarkers source:
- The AUC will be calculated as

AUC (0-Day x) = 
$$\sum_{0-1} \{ \frac{1}{2} (C_i + C_{i+1}) (t_{i+1} - t_i) \}$$

Where,

C<sub>i</sub> = level of biomarker at actual time point i in Day

t<sub>i</sub> = actual time of assessment for time point i in Day

i = actual time of assessment in Day (e.g. Day 1, 3, 5, 8, 16, 24, 32,day 45)

I = last i (Day 5, Day 45, or PT Day 3)

- Actual study day will be used for the AUC calculation.
- When baseline value of a biomarker is missing, AUC for the biomarker will be missing.
- When a subject has only baseline value, AUC will be missing.
- When value of a biomarker is missing between visits, there will be no imputation for the missing value, e.g. subject has day 1, 3, 5, 8, 16, 32, 45 values, and day 24 value is missing, day 24's value will not be imputed, AUC will be calculated using day 1,3,5, 8,16, 32, and 45 values.
- When value of a biomarker is missing at the end, last observation carried forward (LOCF) will be used to impute missing value, e.g, subject has day 1, 3, 5, 8, 16, 24, 32 values and day 45 is missing, day 45 value will be imputed using day 32 value (day 45 value will be assumed the same as day 32 value).
- The value of the AUC(0-45) biomarker is missing if there is no assessment beyond week 24.
- The length of time from Baseline to PT Day 3 visit will vary for subjects who prematurely
  discontinue the study and so the biomarker will also vary.

#### 11.6.6. Health Outcomes

The FLU-PRO Total score is computed as a mean score across all 32 items comprising the instrument. Total scores can range from 0 (symptom free) to 4 (very severe symptoms).

Six domain scores are also computed, representing symptom severity in each of the following body areas: Nose, Throat, Eyes, Chest/Respiratory, Gastrointestinal, and Body/Systemic. Each domain score is calculated as the mean of all items comprising the domain. Each FLU-PRO domain score also ranges from 0 to 4. Algorithms and instructions for computing scores for the FLU-PRO Total and domain scores (including rules for handling missing data) are provided below:

| Domain | Items | Scoring | Minimum Data<br>Requirement |
|---|---|---|---|
| Nose | Runny or dripping nose<br>Congested or stuffy nose<br>Sneezing<br>Sinus pressure | Arithmetic mean of 4 items within <b>Nose</b> domain | 3 of 4 items must<br>be present to<br>calculate domain<br>score |
| Throat | Scratchy or itchy throat<br>Sore or painful throat<br>Difficulty swallowing | Arithmetic mean of 3 items within <b>Throat</b> domain | 2 of 3 items must<br>be present to<br>calculate domain<br>score |
| Eyes | Teary or watery eyes Sore or painful eyes Eyes sensitive to light | Arithmetic mean of 3 items within <b>Eyes</b> domain | 2 of 3 items must<br>be present to<br>calculate domain<br>score |
| Chest/Respiratory | Trouble breathing Chest congestion Chest tightness Dry or hacking cough Wet or loose cough Coughing Coughed up mucus or phlegm | Arithmetic mean of 7 items within Chest/Respiratory domain | 5 of 7 items must<br>be present to<br>calculate domain<br>score |
| Gastrointestinal | Felt nauseous Stomach ache How many times did you vomit? How many times did you have diarrhea? | Arithmetic mean of 4 items within Gastrointestinal domain | 3 of 4 items must<br>be present to<br>calculate domain<br>score |
| Body/Systemic | Headache Head congestion Felt dizzy Lack of appetite Sleeping more than usual Body aches or pains Weak or tired Chills or shivering Felt cold Felt hot Sweating | Arithmetic mean of 11 items within Body/Systemic domain | 8 of 11 items<br>must be present<br>to calculate<br>domain score |

| Total | All above 32 items | Arithmetic mean of all 32 items within FLU-PRO | In the presence of missing data, the above conditions for the calculation of all domain scores must be met in order to calculate the FLU-PRO |
|---|---|---|---|
| | | | total score. |

# 11.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as a subject who completed the Day 45 assessment.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |

#### 11.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will not be<br/>imputed.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events,<br>Exposure | <ul> <li>No missing data is expected for AE and EX.</li> <li>Data Management will query any missing date of AE or EX.</li> </ul> |

### 11.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Time to<br>Clinical<br>Resolution | <ul> <li>For the primary analysis, a Discontinuation=Failure approach will be used (see Section 7.1.2). This approach handles two types of missing data: <ul> <li>due to subjects who prematurely discontinued the study</li> <li>sporadic missing vital sign assessments</li> </ul> </li> </ul> |

# 11.8. Appendix 8: Values of Potential Clinical Importance

## 11.8.1. Laboratory Values

Laboratory parameter will be graded according to the Division of AIDS (DAIDS) toxicity scales (protocol Section 12.5).

#### 11.8.2. ECG

The following subdivision will be used to summarize the absolute and increase from baseline QTc interval data, and absolute PR interval by category

| ECG Parameter | Potential Clinical Importance Range (PCI) | Unit |
|---|---|---|
| Absolute QTc Interval | >450 to ≤480 | msec |
| Absolute QTc Interval | >480 to ≤500 | msec |
| Absolute QTc Interval | >500 | msec |
| Increase from Baseline QTc | >30 to ≤60 | msec |
| Increase from Baseline QTc | >60 | msec |
| Absolute PR interval | 210-250 | msec |
| Absolute PR interval | >250 | msec |

## 11.8.3. Vital Signs

Due to patient population, vital signs will not be flagged as potential clinical importance.

# 11.9. Appendix 9: Examination of Covariates, Subgroups & Other Strata

## 11.9.1. Examination of Covariates, Subgroups & Other Strata

Given the small number of subjects, no subgroups will be assessed.

# 11.10. Appendix 10: Multiple Comparisons & Multiplicity

#### 11.10.1. Handling of Multiple Comparisons & Multiplicity

There will be no adjustments for multiplicity.

# 11.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

### 11.11.1. Statistical Analysis Assumptions

Not applicable

## 11.12. Appendix 12 – Abbreviations & Trade Marks

#### 11.12.1. Abbreviations

#### 11.12.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

**RELENZA** 

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Captisol |
| FluPRO |
| KATZ ADL |
| SAS |
| Tamiflu |

# 11.13. Appendix 13: List of Data Displays

## 11.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacodynamic / Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Pharmacokinetic / Pharmacodynamic | 7.1 to 7.n | 7.1 to 7.n |
| Health Outcome | 8.1 to 8.n | 8.1 to 8.n |
| Virology | 9.1 to 9.n | 9.1 to 9.n |
| Section | List | ings |
| ICH Listings | 1 t | 0 X |
| Other Listings | y t | 0 Z |

# 11.13.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 14: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Biomarker | BM_Fn | BM_Tn | BM_Ln |
| Pharmacodynamic / Biomarker | BMPD_Fn | BMPD_Tn | BMPD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |
| Health Outcomes | HO_Fn | HO_Tn | HO_Ln |
| Virology | VR_Fn | VR_Tn | VR_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 11.13.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|------------------------------------------------|
| DL | Data Look (blinded dry run) |
| IA | Interim Analysis Statistical Analysis Complete |
| HL | Headline |
| SAC | Final Statistical Analysis Complete |

## NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 11.13.4. Study Population Tables

| Study I | Study Population Tables | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| Subjec | t Disposition | | | |
| 1.1. | ITT-E | ES1 | Summary of Subject Disposition | |
| 1.2. | ITT-E | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | |
| Protoc | ol Deviation | | | |
| 1.3. | ITT-E | DV1 | Summary of Important Protocol Deviations | |
| Popula | tion Analysed | | | |
| 1.4. | All Subjects<br>Screened | SP1 | Summary of Study Populations | |
| Demog | raphic and Bas | eline Characteris | tics | |
| 1.5. | ITT-E | DM1 | Summary of Demographic Characteristics | Add age groups <35, 35-<50, >=50 and < 65, >=65.<br>Add BMI and BMI categories <=20, 20-<=25, 25-<br><=30, 30-<=35, 40-<=45,>45. Add tobacco use. |
| 1.6. | ITT-E | DM5 | Summary of Race and Racial Combinations | |
| Prior a | Prior and Concomitant Medications | | | |
| 1.7. | ITT-E | POP T2 | Summary of Prior Exposure to Oseltamivir | Add a footnote "Only influenza therapies taken within 7 days of baseline visit were collected" CMPRIOR='Y'' or if medication started prior to IP start.No imputation for missing values |

| Study F | Study Population Tables | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| 1.8. | ITT-E | CM1 | Summary of Prior Anti-influenzaTherapy | Includes pre-treatment CMs used for Anti-influenza therapy. Study team to review & provide list of CM terms prior to DBR Add a footnote "Only influenza therapies taken within 7 days of baseline visit were collected" |
| | | | | Consider post-treatment as those records where the |
| 1.9. | ITT-E | CM1 | Summary of Post-Treatment Anti-influenzaTherapy | conmed start or end date are after the IP end date. Apply same logic for Table 1.11 |
| | | | | Add a column for "Pre-Treatment Steriod Use" |
| | | | | Add a footnote "Only influenza therapies taken within 7 days of baseline visit were collected" |
| 1.10. | D. ITT-E CM1 | | Summary of Pre-Treatment Steroids Use by Duration of Time | the steroid use will be grouped as 3 categories, <1 week, 1 week - <6 months and 6 months and more, the table will summarize the number and percent of subject in each group |
| 1.11. | ITT-E | CM1 | Summary of Post-Treatment Steroid Use | |
| Other | • | | | |
| 1.12. | ITT-E | POP T3 | Summary of Flu Type and Symptoms | Includes influenza subtypes |
| 1.13. | ITT-E | MH4 | Summary of Past and Current Medical Conditions | By 'Past', 'Current', 'No' |
| 1.14. | ITT-E | POP T4 | Summary of Ventilation Status at Baseline | |
| 1.15. | ITT-E | POP T6 | Summary of Exposure to Study Treatment | |
| 1.16. | IPP | POP T4 | Summary of Ventilation Status at Baseline | |

# 11.13.5. Efficacy Tables

| Efficacy Tables | | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes |
| Efficacy | | | | |
| 2.1. | IPP | EFF T2 | Summary of Improved Clinical Response | |
| 2.2. | IPP | EFF T6 | Summary of Improved Respiratory Response | |
| 2.3. | IPP | | Summary of Post Baseline Ventilation Status | Mock per IVZ |
| 2.4. | IPP | CM1 | Summary of Frequency of Associated Antibiotic Use for Treatment of Complications of Influenza | List will be identified by study team prior to unblinding |

# 11.13.6. Efficacy Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 2.1. | IPP | EFF F1 | Individual Plot of Time to Clinical Response | 10 lines for 10 subjects with different symbols representing event or censoring and different color representing different treatment. |


| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 2.2. | IPP | EFF F1 | Individual of Time to Respiratory Response (Improved Respiratory Status) | 10 lines for 10 subjects with different symbols representing event or censoring and different color representing different treatment, including any subject who resolved prior to baseline (negative response time, with a footnote). |

# 11.13.7. Safety Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 3.1. | Safety | SAFE T1 | Summary of All Adverse Events by System Organ Class and Maximum Grade | Please add a footnote to indicate "Mild or Grade 1", "Moderate or Grade 2", "Severe or Grade 3", "Grade 4". |
| 3.2. | Safety | AE3 | Summary of All Adverse Events by Overall Frequency | |
| 3.3. | Safety | AE3 | Summary of Grade 2-4 Adverse Events by Overall Frequency | |
| 3.4. | Safety | AE3 | Summary All Drug-Related Adverse Events by Overall Frequency | |
| 3.5. | Safety | AE1 | All Non-Serious Adverse Events by SOC and PT | Eudra |
| 3.6. | Safety | AE16 | SAE with number of subjects and number of occurrences by SOC and PT | Eudra |
| 3.7. | Safety | AE3 | Summary of Drug-Related Grade 2-4 Adverse Events by Overall Frequency | |
| 3.8. | Safety | AE3 | Summary of Adverse Events of Special Interest by Overall Frequency | AE terms for AESI will be provided prior to unblinding. |
| 3.9. | Safety | AE8 | Listing of Adverse Events for Subjects with Neutropenia (>= Grade 1) | |
| 3.10 | ). Safety | AE3 | Summary of Non-Fatal Serious Adverse Events | |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 3.1 | 1. Safety | AE1 | Summary of Serious Adverse Events by System Organ Class | |
| 3.1 | 2. Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class | |
| 3.1 | 3. Safety | AE3 | Summary of Drug-Related Non-Fatal Serious Adverse Events | |
| 3.1 | 4. Safety | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | |
| 3.1 | 5. Safety | | Summary of Maximum Treatment Emergent Toxicities of All Lab Parameters | IDMC output |
| 3.1 | 6. Safety | SAFE T2 | Summary of Data Supporting Safety Halting Criteria | |
| 3.1 | 7. Safety | LB1 | Summary of Creatinine by Visit | |
| 3.1 | Safety<br>8. | LB1 | Summary of Change from Baseline for Serum WBCs, %<br>Neutrophils, and Absolute Neutrophils Counts, Creatinine, Liver<br>Function Test | IDMC output |
| 3.1 | 9. Safety | LB1 | Summary of Absolute Neutrophils Count by Visit | |

# 11.13.8. Safety Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 3.1. | Safety | | Individual Plot of Creatinine by Visit by Subject | |
| 3.2. | Safety | | Individual Plot of Absolute Neutrophils Count by Visit by Subject | Page per each subject with a vertical line on day of treatment discontinued, include treatment, sex, age, in addition to subject ID |

## 11.13.9. Pharmacokinetic Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 4.3 | PK | PK06 | Summary of Derived Whole Blood Danirixin PK Parameters (non-transformed and log-transformed) by Treatment | |
| 4.4 | PK | PK01 | Summary of Whole Blood Danirixin Pharmacokinetic<br>Concentration-Time Data (insert units) by Treatment and<br>Day | Replace (insert units) with unit of measure. Include all subjects |

# 11.13.10. Pharmacokinetic Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 4.1 | PK | PK20 | Median (IR) Plot of Whole Blood Danirixin Concentration-<br>Time Plot (Linear and Semi-Log) by Treatment | Include line for LLQ along with footnote defining LLQ value Overlay Day 1, 3 and 5. |
| 4.2 | PK | PK20 | Mean (SE) Plot of Whole Blood Danirixin Concentration-<br>Time Plot (Linear and Semi-Log) by Treatment | Include line for LLQ along with footnote defining LLQ value Overlay Day 1, 3 and 5. |
| 4.5 | PK | PK16a | Individual Whole Blood Danirixin Concentration-Time Plots by Subject (Linear and Semi-log) | 1. X-axis displays actual relative time 2. Include line for LLQ along with footnote defining LLQ value 3. Include values below LLQ 4. Overlay Day 1, 3 and 5 |

# 11.13.11. Biomarker Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 5.1. | IPP | BM_F2 | Individual Plot of Serum Biomarkers by Visit by Subject - Influenza Positive Population | spaghetti plot, one plot per biomarker<br>per matrix. Subject ID and treatment<br>group should be identifiable by<br>color/symbol |
| 5.2. | IPP | BM_F2 | Individual Plot of Nasal Wash Biomarkers by Visit by Subject - Influenza Positive Population | spaghetti plot, one plot per biomarker.<br>Subject ID and treatment group should<br>be identifiable by color/symbol |


| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 5.3. | IPP | BM_F2 | Individual Plot of Nasal SAM Strips Biomarkers by Visit by Subject - Influenza Positive Population | spaghetti plot, one plot per biomarker.<br>Subject ID and treatment group should<br>be identifiable by color/symbol |
| 5.4. | IPP | BM_F2 | Individual Plot of BAL Biomarkers by Visit by Subject - Influenza Positive Population | spaghetti plot, one plot per biomarker.<br>Subject ID and treatment group should<br>be identifiable by color/symbol |

# 11.13.12. Pharmacodynamic / Biomarker Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 6.1. | IPP | BMPD_F3 | Matrix Comparative Plot of Individual Scatter Plot of Biomarkers vs Biomarkers for Each Biomarker Source by Select Visits | One page per biomarker. The x on y axis will contain the 5 biomarkers: Serum, Nasal wash, Nasal SAM Strips, BAL Include the pearson's correlation coefficient and p-value on the graph. Use one color One page for Day 1, Day 5, Day 45, PT Day 3 |
| 6.2. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Serum<br>Biomarkers vs. Time to Clinical Response - Influenza<br>Positive Population | One page per biomarker. TTCR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTCR, AUC(0-45) vs TTCR, AUC(0-PT Day 3) vs TTCR, Different color for treatment. Include a regression line for each treatment group |
| 6.3. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Serum Biomarkers vs. Time to Respiratory Response - Influenza Positive Population | One page per biomarker. TTRR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTRR, AUC(0-45) vs TTRR, AUC(0-PT Day 3) vs TTRR, Different color for treatment. Include a regression line for each treatment group |
| 6.4. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Nasal<br>Wash Biomarkers vs. Time to Clinical Response -<br>Influenza Positive Population | One page per biomarker. TTCR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTCR, AUC(0-45) vs TTCR, AUC(0-PT Day 3) vs TTCR, Different color for treatment. Include a regression line for each treatment group |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 6.5. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Nasal<br>Wash Biomarkers vs. Time to Respiratory Response -<br>Influenza Positive Population | One page per biomarker. TTRR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTRR, AUC(0-45) vs TTRR, AUC(0-PT Day 3) vs TTRR, Different color for treatment. Include a regression line for each treatment group |
| 6.6. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Nasal SAM Strips Biomarkers vs. Time to Clinical Response - Influenza Positive Population | One page per biomarker. TTCR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTCR, AUC(0-45) vs TTCR, AUC(0-PT Day 3) vs TTCR, Different color for treatment. Include a regression line for each treatment group |
| 6.7. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve Nasal SAM Strips Biomarkers vs. Time to Respiratory Response - Influenza Positive Population | One page per biomarker. TTRR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTRR, AUC(0-45) vs TTRR, AUC(0-PT Day 3) vs TTRR, Different color for treatment. Include a regression line for each treatment group |
| 6.8. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve BAL<br>Biomarkers vs. Time to Clinical Response - Influenza<br>Positive Population | One page per biomarker. TTCR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTCR, AUC(0-45) vs TTCR, AUC(0-PT Day 3) vs TTCR, Different color for treatment. Include a regression line for each treatment group |
| 6.9. | IPP | BMPD_F1 | Individual Scatter Plot of Area Under the Curve BAL Biomarkers vs. Time to Respiratory Response - Influenza Positive Population | One page per biomarker. TTRR on y axis, AUC biomarker on x axis. AUC(0-5) vs TTRR, AUC(0-45) vs TTRR, AUC(0-PT Day 3) vs TTRR, Different color for treatment. Include a regression line for each treatment group |

# 11.13.13. Pharmacokinetic / Pharmacodynamic Tables

Not Applicable

# 11.13.14. Pharmacokinetic / Pharmacodynamic Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 7.12 | IPP | | Target Engagement Biomarker versus DNX PK Parameters | Target engagement biomarkers include IL-8, MPO, neutrophil elastase and neutrophil counts (the one from nasal wash, not the one from blood) |

## 11.13.15. Health Outcome Tables

| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 8.1. | IPP | HO T2 | Summary of Change from Baseline in KATZ ADL Score and each ADL Activity | Includes baseline value |
| 8.2. | IPP | HO T5 | Summary of FLU-PRO Total and Domain Scores | Use "Baseline" for label instead of<br>"Baseline for CFB" |
| 8.3. | IPP | HO T5 | Summary of Change from Baseline FLU-PRO Total and Domain Scores | Includes baseline value |

# 11.13.16. Virology Tables

| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 9.1. | IPP | VR T1 | Summary of Change from Baseline in Influenza Viral Load by qRT-PCR (log 10 VP/mL) Overall | Includes baseline value<br>Summarize by A and B combined |
| 9.2. | IPP | VR T2 | Summary of Change from Baseline in Influenza Viral Load by qVC (log10 TCID50/mL) for Subjects Culture Positive at Baseline –Nasopharyngeal | Includes baseline value |
| 9.3. | ITTE | VR T7 | Proportion of Subjects with Other Co-infected Viruses by Multiplex RT PCR. | |
| 9.4. | IPP | VR T4 | Summary of Resistance Associated Mutations Detected in the NA Gene by Subtype - Nasopharyngeal | |
| 9.5. | IPP | VR T4 | Summary of Resistance Associated Mutations Detected in the HA Gene by Subtype - Nasopharyngeal | |

# 11.13.17. Virology Figures

| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
|---|---|---|---|---|
| 9.1. | IPP | VR F1 | Individual Plot of Change from Baseline in Influenza Viral Load by qRT-PCR (log10 VP/mL) by Subject for Influenza A and B - Nasopharyngeal | Include zero at baseline |
| 9.2. | IPP | VR F1 | Individual Plot of Change from Baseline in Influenza Viral Load by qVC (log10 TCID50/mL) for Subjects Culture Positive at Baseline -Nasopharyngeal | Include zero at baseline |

# 11.13.18. ICH Listings

| ICH : Li | ICH : Listings | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| Subjec | Disposition | | | |
| 1. | All Subjects<br>Screened | ES7 | Listing of Screen Reasons for Screen Failure | |
| 2. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | |
| 3. | ITT-E | SD2 | Listing of Reasons for Study Treatment Discontinuation | |
| 4. | ITT-E | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | |
| 5. | ITT-E | TA1 | Listing of Planned and Actual Treatments | |
| Protoco | ol Deviations | | | |
| 6. | ITT-E | DV2 | Listing of Important Protocol Deviations | |
| 7. | ITT-E | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | |
| Popula | tions Analysed | | | |
| 8. | All Subjects<br>Screened | SA3a | Listing of Subjects Excluded from Any Population | |
| Demog | Demographic and Baseline Characteristics | | | |
| 9. | ITT-E | DM2 | Listing of Demographic Characteristics | |
| 10. | ITT-E | DM9 | Listing of Race | |

| ICH : Li | ICH : Listings | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| 11. | ITT-E | CM2 | Listing of Concomitant Medications | Add column to indicate 'complications of influenza' |
| 12. | ITT-E | MH2 | Listing of Past and Current Medical Conditions | |
| 13. | ITT-E | MH2 | Listing of Subjects with Renal Impairment | Renal impairment is based on Creatinine Clearance Criteria Any time during study including baseline and post baseline |
| 14. | IIT-E | CM2 | Listing of Subjects with Prior Oseltamivir Exposure | |
| Exposu | re and Treatme | ent Compliance | | |
| 15. | Safety | EX3 | Listing of Exposure Data | |
| Advers | e Events | | | |
| 16. | Safety | AE8 | Listing of All Adverse Events | Add asterisk for subjects with baseline renal impairment |
| 17. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | |
| 18. | Safety | AE8 | Listing of Adverse Events of Special Interest | |
| Serious | and Other Sig | nificant Adverse l | Events | |
| 19. | Safety | AE8 | Listing of Fatal Adverse Events | |
| 20. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | |
| 21. | Safety | SAFE L1 | Listing of Reasons for Considering as a Serious Adverse Event | Use study 201682 as a reference |

| ICH : Li | ICH : Listings | | | |
|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| 22. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | |
| 23. | Safety | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment` | |
| 24. | Safety | MH2 | Listing of Subjects with Liver Stopping Events | |
| All Lab | oratory | | | |
| 25. | Safety | LB5 | Listing of Laboratory Data for Subjects with Abnormalities of Potential Clinical Concern (Grade 3-4) | |
| 26. | Safety | LB5 | Listing of All Laboratory Data | |
| ECG | | | | |
| 27. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with a Value of Potential Clinical Importance | |
| 28. | Safety | CP_EG5 | Listing of Abnormal ECG Findings | |

# 11.13.19. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Need for early<br>terminated<br>study |
| Popula | ition | | | | |
| 29. | ITT-E | POP L1 | Listing of Flu Type and Symptoms | | |
| 30. | ITT-E | POP L2 | Listing of Chest X-Ray Results | Indicate if subject is included | d in IPP |
| Efficacy | у | | | | |
| 31. | IPP | EFF L1 | Listing of Time to Clinical Response | | |
| 32. | IPP | EFF L2 | Listing of Time to Respiratory Response | | |
| 33. | IPP | | Listing of Vital Signs | | |
| 34. | IPP | | Listing of Ventilation Status – Mechanical Ventilation | Use NAI114373 as a refer<br>Add start and stop time | |
| 35. | IPP | | Listing of Ventilation Status – Supplemental Oxygen | Use NAI114373 as a refer Oxygen saturation history should be inc | |
| 36. | IPP | | Listing of Hospital Discharge | Include date, duration and r | reason |
| 37. | IPP | | Listing of Subjects Who Were Admitted to Intensive Care Unit | | |
| Safety | Safety | | | | |
| 38. | Safety | LB5 | Listing of Absolute Neutrophils for Subjects with Grade 3-4 Absolute Neutrophils or AE of Neutropenia | | |
| 39. | Safety | LB5 | Listing of Creatinine for Subjects with Creatinine Increase > 0.5 mg/dl in Two Consecutive Visits | | |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Need for early<br>terminated<br>study |
| PK | | | | | |
| 40. | PK | PK L1 | Listing of Whole Blood Danirixin Pharmacokinetic Concentration Data | Include NQ values | |
| 41. | PK | LPK2 | Listing of Whole Blood Danirixin Derived Pharmacokinetic Parameters | | |
| Biomar | ker | | | | |
| 42. | ITT-E | | Listing of Serum Biomarkers | | |
| 43. | ITT-E | | Listing of Nasal Wash Biomarkers | | |
| 44. | ITT-E | | Listing of Nasal SAM Strips Biomarkers | | |
| 45. | ITT-E | | Listing of BAL Biomarker | | |
| Virolog | У | | | | |
| 46. | ITT-E | VR L1 | Listing of Influenza Viral RNA (qRT-PCR and TCID50) in Nasopharyngeal | Use study 201682 as a refe | erence |
| 47. | IPP | VR L2 | Listing of Co-infected Subjects | | |
| 48. | ITT-E | | Listing of Other Viruses by Multiplex RT PCR. | | |
| 49. | ITT-E | | Listing of Phenotypic IC50 Results | Use NAI114373 as a refer | ence |
| 50. | IPP | | Listing of Resistant Mutations in NA and HA Genes | Use NAI114373 as a refer | ence |
| Health | Outcome | | | , | |
| 51. | IPP | HO L1 | Listing of Hospital Readmission | | |
| 52. | IPP | HO L2 | Listing of ADL KATZ Score and each ADL Activity | | |
| 53. | IPP | HO L3 | Listing of 3-Point Scale (Bed Rest, Limit Ambulation, Unrestricted) | | |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Need for early<br>terminated<br>study |
| 54. | IPP | HO L4 | Listing of FLU-PRO Total and Domain Scores | | |

# 11.14. Appendix 14: Example Mock Shells for Data Displays

The mock shells for data displays are contained in a separate document.